CLINICAL TRIAL: NCT04728204
Title: Internet-based Cognitive Behavioral Therapy for Depressed Elderly: a Two-armed Randomized Controlled Trial
Brief Title: Internet-based Psychotherapy for Depressed Elderly
Acronym: iPSYDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Jonas Eimontas, Associate Professor, Senior Research Fellow, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iPSYDE_1_2021
Record Dates: First submitted 2021-01-15; First posted 2021-01-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Depression
Keywords: Depression; Internet-based cognitive behaviour therapy; Elderly; eHealth
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either control or intervention group. Participants in the control group will receive the same treatment after the intervention group is finished with the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): 8 module, 8 week long internet-based intervention for reducing burden of depression
  Interventions: Behavioral: Depresijos terapija
- Control group (No Intervention): Participants randomized to the control group will be instructed to wait until the intervention group finishes the treatment and that they will be able to use the same intervention afterwards.

INTERVENTIONS:
Behavioral: Depresijos terapija — Intervention is based on the principles of cognitive behavioral therapy and culturally adapted to elderly Lithuanian population. The main purpose of the intervention is to reduce the symptoms of depression and increase psychological well-being. Intervention contains psychoeducation, examples, exercises and consultation with a psychologist.
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the effectiveness of internet-based cognitive behavioral therapy (CBT) for depressed elderly.

DETAILED DESCRIPTION:
Individuals of age 60+ with symptoms of depression will be assessed before the study. At week 0, participants who meet eligibility requirements will be randomized either to intervention group which will participate in an 8-week internet-based modular CBT or to a delayed treatment control group.

ELIGIBILITY:
Inclusion Criteria:

* depressive symptoms
* have access to a computer/tablet/smartphone and to the internet
* have good knowledge of the Lithuanian language

Exclusion Criteria:

* alcohol addiction
* presently in any other psychological treatment
* severe depression
* suicidal ideation
* significant change in psychiatric medication (during last 6 weeks)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Pre-treatment, week 8, 3, 12 and 24 months post-treatment
  Change from baseline in depression symptoms post-treatment (week 8), at three months, at 12 months and at 24 months post-treatment. Measure contains 9 questions that have to be responded to by choosing an answer from a 4-item Likert scale, where number 0 indicates 'Not at all' and 3 - 'Nearly every day'. Higher score indicates more severe symptoms.
Geriatric Depression Scale (GDS) | Pre-treatment, week 8, 3, 12 and 24 months post-treatment
  Change from baseline in depression symptoms post-treatment (week 8), at three months, at 12 months and at 24 months post-treatment. Measure contains 15 questions that have to be responded 'Yes' or 'No'. Higher score indicates more severe symptoms.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Pre-treatment, week 8, 3, 12 and 24 months post-treatment
  Change from baseline in anxiety symptoms post-treatment (week 8), at three months, at 12 months and at 24 months post-treatment. Measure contains 7 questions that have to be responded to by choosing an answer from a 4-item Likert scale, where number 0 indicates 'Not at all' and 3 - 'Nearly every day'. Higher score indicates more severe symptoms.
The World Health Organisation- Five Well-Being Index (WHO-5) | Pre-treatment, week 8, 3, 12 and 24 months post-treatment
  Change from baseline in well-being post-treatment (week 8), at three months, at 12 months and at 24 months post-treatment. WHO-5 contains 5 statements about individuals well-being in the past two weeks. Respondents have to choose the best corresponding answer using a 6-item Likert scale where a score of 0 indicates 'At no time' and a score of 5 - 'All the time'. Higher score indicates higher well-being.

OTHER OUTCOMES:
The Alcohol Use Disorders Identification Test (AUDIT) | Pre-treatment
  AUDIT will be used for alcohol consumption and related risks assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Eimontas, PhD, Principal Investigator — Vilnius University
Locations (1):
- Vilnius University, Vilnius, Lithuania, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eimontas J, Pakalniskiene V, Biliunaite I, Andersson G. A tailored Internet-delivered modular intervention based on cognitive behavioral therapy for depressed older adults: a study protocol for a randomized controlled trial. Trials. 2021 Dec 16;22(1):925. doi: 10.1186/s13063-021-05903-4. PMID 34915909